CLINICAL TRIAL: NCT02975791
Title: Ultrasonography Versus Palpation for Identification of the Cricothyroid Membrane
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Seltz Kristensen, Consultant, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Ultrasound MC 24112016
Record Dates: First submitted 2016-11-20; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Airway Obstruction
Keywords: Airway Obstruction
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- palpation (Active Comparator): Marking the cricothyroid membrane after ultrasound
  The intervention is to mark the cricothyroid membrane in order to know exactly where it is in case that it should be needed fur emergency cricothyrotomy. The doctors mark the cricothyroid membrane with a pen after using palpation for identification.
  Interventions: Procedure: Marking of the cricothyroid membrane after Palpation
- ultrasound (Active Comparator): Marking of the cricothyroid membrane after Palpation
  intervention is to mark the cricothyroid membrane in order to know exactly where it is in case that it should be needed fur emergency cricothyrotomy doctors mark the cricothyroid membrane with a pen after using ultrasonography for the identification
  Interventions: Other: Marking the cricothyroid membrane after ultrasound

INTERVENTIONS:
Other: Marking the cricothyroid membrane after ultrasound — Ultrasonography is applied to the subjects neck in order to identify the cricothyroid membrane - subsequently the membrane is marked with a pen
  Arms: ultrasound
Procedure: Marking of the cricothyroid membrane after Palpation — Palpation is applied to the subjects neck in order to identify the cricothyroid membrane- subsequently the membrane is marked with a pen
  Arms: palpation

SUMMARY:
After a structured teaching program anaesthetists are educated in identifying the cricothyroid membrane with ultrasonography. Thereafter their ability to do so is compared with their ability to do so with palpation. In an obese volunteer

DETAILED DESCRIPTION:
After a structured teaching program anaesthetists are educated in identifying the cricothyroid membrane with ultrasonography. Thereafter their ability to do so is compared with their ability to do so with palpation.

The purpose is to advise a propriety method for preanesthetic identification. In an obese volunteer

ELIGIBILITY:
Inclusion Criteria:

* BMI > 40
* Female

Exclusion Criteria:

* Age below 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Frequency of correct identification of the cricothyroid membrane | "2 min"
  The fraction of cases where the cricothyroid membrane is identified correctly

SECONDARY OUTCOMES:
time to correct identification of the cricothyroid membrane | "2 min"
  The time consumed for correct identification of the cricothyroid membrane

IPD SHARING:
Plan to Share IPD: No